CLINICAL TRIAL: NCT01130025
Title: Efficacy and Safety of Long-Term (6 Months) Innohep® Treatment Versus Anticoagulation With a Vitamin K Antagonist (Warfarin) for the Treatment of Acute Venous Thromboembolism in Cancer Patients / IN 0901 INT
Brief Title: Long-Term Innohep® Treatment Versus a Vitamin K Antagonist (Warfarin) for the Treatment of Venous Thromboembolism (VTE) in Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN 0901 INT; 2009-018141-20 (EudraCT Number)
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2014-06

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Warfarin; Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Innohep® (Experimental): Long-term treatment with Innohep® only.
  Interventions: Drug: Innohep®
- Warfarin (Active Comparator): Oral treatment with warfarin in combination with overlapping initial (5 to 10 days) treatment with Innohep®.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Tablets. Once daily for 6 months (180 days) to maintain therapeutic international normalised ratio (INR) levels in combination with initial (5-10 days) overlapping treatment with Innohep®.
  Arms: Warfarin
Drug: Innohep® — Solution for sub-cutaneous injection, pre-filled syringes. Once daily for 6 months (180 days). 175 anti Xa IU/kg.
  Arms: Innohep®

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Innohep® in preventing the recurrence of VTE in patients with active cancer who have had an acute VTE episode.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of active cancer.
* Symptomatic and objectively confirmed VTE.
* ≥ 18 years of age or above the legal age of consent as per country specific regulations.
* Patients with Eastern Co-operative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Signed informed consent.

Exclusion Criteria:

* Life expectancy < 6 months.
* Patients with basal cell carcinoma or non-melanoma skin cancer.
* Creatinine clearance ≤ 20 ml/min.
* Contra-indications to anticoagulation.
* Known hypersensitivity to the investigational product (Innohep®) or the reference product (warfarin).
* History of heparin-induced thrombocytopenia (HIT).
* Pre-randomisation therapeutic anticoagulant treatment for acute VTE administered for more than 72 hours prior to randomisation.
* Patients unlikely to comply with the protocol.
* Participation in another interventional study.
* Pregnant or breast-feeding women.
* Women of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Composite end-point represented by the time in days from randomisation to the first occurrence of VTE | 6 months
  * Symptomatic non-fatal DVTs.
  * Symptomatic non-fatal PEs.
  * Fatal PE.
  * Incidental proximal DVT (popliteal vein or higher).
  * Incidental proximal PE (segmental arteries or larger).

SECONDARY OUTCOMES:
Time in days from randomisation to the first occurrence of VTE. | 6 months
  * The 5 individual components of the composite primary efficacy endpoint.
  * A composite endpoint of symptomatic DVT and/or PE, including fatal PE.
  Safety endpoints will consist of bleeding and overall mortality

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Y. Y. Lee, MD, MSc, FRCPC, Principal Investigator — Director of Thrombosis, Division of Hematology, University of British Columbia, Canada
Locations (1):
- Diamond Health Care Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kahale LA, Matar CF, Hakoum MB, Tsolakian IG, Yosuico VE, Terrenato I, Sperati F, Barba M, Schunemann H, Akl EA. Anticoagulation for the initial treatment of venous thromboembolism in people with cancer. Cochrane Database Syst Rev. 2021 Dec 8;12(12):CD006649. doi: 10.1002/14651858.CD006649.pub8. PMID 34878173
- [Derived] Bauersachs R, Lee AYY, Kamphuisen PW, Meyer G, Janas MS, Jarner MF, Khorana AA; CATCH Investigators. Renal Impairment, Recurrent Venous Thromboembolism and Bleeding in Cancer Patients with Acute Venous Thromboembolism-Analysis of the CATCH Study. Thromb Haemost. 2018 May;118(5):914-921. doi: 10.1055/s-0038-1641150. Epub 2018 Apr 4. PMID 29618162
- [Derived] Lee AYY, Kamphuisen PW, Meyer G, Bauersachs R, Janas MS, Jarner MF, Khorana AA; CATCH Investigators. Tinzaparin vs Warfarin for Treatment of Acute Venous Thromboembolism in Patients With Active Cancer: A Randomized Clinical Trial. JAMA. 2015 Aug 18;314(7):677-686. doi: 10.1001/jama.2015.9243. PMID 26284719
- [Derived] Lee AY, Bauersachs R, Janas MS, Jarner MF, Kamphuisen PW, Meyer G, Khorana AA; CATCH Investigators. CATCH: a randomised clinical trial comparing long-term tinzaparin versus warfarin for treatment of acute venous thromboembolism in cancer patients. BMC Cancer. 2013 Jun 13;13:284. doi: 10.1186/1471-2407-13-284. PMID 23764005